CLINICAL TRIAL: NCT01944462
Title: Impact and Cost of a Pharmacist Pneumococcal Vaccination Program With PNEUMOVAX® 23 at an Urban Senior Center for Adults Aged 65 Years or Older or Those With Defined Risk Factors for Invasive Pneumococcal Disease
Brief Title: Impact and Cost of a Pharmacist Pneumococcal Vaccination Program With PNEUMOVAX® 23 at an Urban Senior Center
Acronym: PPVP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Merck IISP ID 50926
Record Dates: First submitted 2013-09-05; First posted 2013-09-17 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-05

CONDITIONS: Study is Open to Seniors Age 50 or Older
Keywords: pneumococcal vaccine; pharmacist vaccination; Pneumovax 23; pneumococcal vaccine polyvalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacist Pneumococcal Vaccine Program (PPVP) (Experimental): Individuals receiving the PPVP intervention which consists of the educational program delivered on site at the collaborating senior center.
  Interventions: Behavioral: Pharmacist Pneumococcal Vaccine Program (PPVP)

INTERVENTIONS:
Behavioral: Pharmacist Pneumococcal Vaccine Program (PPVP) — 1.5 hour educational intervention delivered onsite at collaborating senior center consisting of 3 components: presentation about pneumococcal disease and the vaccine given by a infectious disease-certified pharmacist; 2) skits given by volunteer actors at the senior center to illustrate real world scenarios related to pneumococcal disease and the vaccine; 3) action planning to consist of small group breakouts led by licensed pharmacists and 4) vaccination day which is an optional component following the education program, for participants eligible to receive the vaccine. Vaccination to be provided free of charge to eligible participants who opt to receive it.

SUMMARY:
The overall goals of this program are to measure the impact of a pharmacist pneumococcal vaccine education program (PPVP) using a senior center model of care and provide the pneumococcal vaccine to eligible participants.

Hypotheses

1. PPVP will result in improved knowledge and awareness in older minorities in the senior center setting (primary hypothesis);
2. Participants who are vaccinated through the project will experienced increased trust in receiving vaccines from a pharmacist;
3. Participants will be satisfied with and trust the PV information provided by pharmacists in the PPVP;
4. PPVP is an efficient approach to educating patients in the senior center based on its costs;
5. Participating pharmacists will be activated to implement PPVP learnings in their practice.

ELIGIBILITY:
Inclusion Criteria:

A. Inclusions for PPVP:

1. Age ≥ 50 years old
2. Can attend a 1.5-hour session at CIP
3. Cognitively intact based on responses to an Abbreviated Mental Test Score (AMTS) of ≥7 (see Appendix for AMTS instrument)
4. Can speak and read English at ≥4th grade level as evidenced by ability to read a brief passage
5. Access to a telephone

B. Inclusions to receive the optional pneumococcal vaccination:

Patient meets ≥1 of the following criteria for receiving their first pneumococcal vaccination:

1. All adults age 65 years and older who have not had the vaccine previously
2. Age 50-64 years with any of the following conditions:

   1. Cigarette smokers age 19 years and older
   2. Chronic cardiovascular disease (e.g., congestive heart failure, cardiomyopathies; excluding hypertension)
   3. Chronic pulmonary disease (including COPD and emphysema, and for adults ages 19 years and older, asthma)
   4. Diabetes mellitus
   5. Alcoholism
   6. Chronic liver disease, cirrhosis
   7. Candidate for or recipient of cochlear implant
   8. Functional or anatomic asplenia (e.g., sickle cell disease, splenectomy)
   9. Immunocompromising conditions or on immunosuppressive therapy
   10. Chronic renal failure or nephrotic syndrome

OR

Patient meets ≥1 of the following criteria for receiving a booster dose of the pneumococcal vaccination:

1. Adults age 65 years and older who received their first dose for any indication when they were younger than age 65 years.
2. Adults age 50-64 who have not received the vaccine for ≥5 years and have one of the following conditions:

   1. Functional or anatomic asplenia (including persons with sickle cell disease or splenectomy patients);
   2. Chronic renal failure (including dialysis patients) or nephrotic syndrome;
   3. Immunocompromising conditions or on immunosuppressive therapy

Exclusion Criteria:

A. Exclusions to the PPVP program: none

B. Exclusions to receiving the optional pneumococcal vaccine:

1. Participant has a history of allergic reaction to pneumococcal vaccine
2. Participant has a history of allergic reaction to any component of any vaccine
3. Participant with moderate or severe illness (these individuals will be advised to speak to their doctor regarding the vaccine)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pizzi, PharmD, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Center in the Park, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and program coordination were completed from January to November 2014, through partnerships with local churches and senior centers.
Pre-assignment Details: Pre/post design (no groups). Inclusion criteria were age ≥50; able to attend a 1.5-hour session; cognitively intact (abbreviated mental test score ≥7); speak & read English at ≥4th grade (ability to read a brief passage). Additionally, program attendees wishing to participate in the study signed consent forms prior to the start of the program.
Groups:
- PPPP Participants: One group (pre/post design) receiving the PPPP intervention
Period: PPPP Educational Program
Arm/Group | PPPP Participants
Started | 203
Baseline | 203
Post-Test | 187
3 Month Follow-Up | 143
Completed | 143
Not Completed | 60
Not completed — Lost to Follow-up | 60
Period: Optional Vaccination
Arm/Group | PPPP Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PPPP Participants
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (8.955)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender, customized: Female | 152
  Gender, customized: Male | 23
  Gender, customized: No response / prefer not to answer | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 163
  White | 2
  More than one race | 0
  Unknown or Not Reported | 38
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: Knowledge and Awareness of Pneumococcal Disease
Description: Change in knowledge and awareness of pneumococcal disease over time were assessed for the following domains: susceptibility to infection, symptoms of disease, severity of illness, and vaccination with an emphasis on vaccine efficacy, safety, and eligibility. Assessments at baseline, post-test (immediately following intervention), and 3 months using the Pneumonia Knowledge Questionnaire, an instrument developed by investigators to assess participants' knowledge and awareness in the domains of interest. Instrument consists of 5 "mark all that apply" items and one "mark the best response" item. Scores range from 0 (no correct responses) to 28 (all responses correct), with a higher score value corresponding to better knowledge and awareness.
Time Frame: Baseline, post-test, 3 months
Population: Intention-to-treat (ITT) sample
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PPPP Participants
Number analyzed (Participants) | 190
scores on a scale
  Baseline knowledge score (max score 28) | 13.90 (6.725)
  Post-test knowledge score (max score 28) | 20.41 (6.254)
  3 month knowledge score (max score 28) | 21.43 (4.524)

2. Secondary Outcome: Trust in Pharmacists as Vaccine Providers
Description: Trust in pharmacists as vaccine providers were measured by comparing responses to the trust items in the baseline, post-test (immediately following intervention), and 3-month assessments. Trust items were coded on a 4-level Likert scale, with lower values corresponding to higher agreement with the trust statements (therefore a lower mean response indicates greater trust). Minimum possible score was 1 (indicating complete trust in pharmacists as vaccine providers) and maximum possible score was 4 (indicating complete lack of trust in pharmacists as vaccine providers).
Time Frame: Baseline, post-test (immediately following intervention), 3 months
Population: Intention-to-Treat (ITT) sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPPP Participants
Number analyzed (Participants) | 190
units on a scale
  Baseline | 1.79 (0.51)
  Post-Test | 1.55 (0.47)
  3 Months | 1.80 (0.43)

3. Secondary Outcome: Activation
Description: Activation was measured as number of participants having taken action at 3 months or planning action at baseline, post-test, and 3 months.
Time Frame: 3 months
Population: Intention-to-Treat (ITT) sample, subset not reporting positive history of pneumococcal vaccination at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PPPP Participants
Number analyzed (Participants) | 113
Participants
  Actions taken at 3 months | 77
  Actions planned at baseline | 41
  Actions planned at post-test | 91
  Actions planned at 3 months | 27

4. Secondary Outcome: Satisfaction With PPPP
Description: Satisfaction with PPPP was measured as participants' overall satisfaction with the content of PPPP, extent to which the participant felt engaged, and belief that the program helped them learn about pneumonia and the vaccination.
Time Frame: 3 months
Population: Intention-to-treat (ITT) sample
Measure: Count of Participants; unit: Participants
Arm/Group | PPPP Participants
Number analyzed (Participants) | 190
Participants
  Satisfied with content: Completely Agree | 69
  Satisfied with content: Somewhat agree | 3
  Satisfied with content: Somewhat disagree | 1
  Satisfied with content: Completely disagree | 1
  Satisfied with content: No response | 116
  Engaged or interested in the program: Completely Agree | 70
  Engaged or interested in the program: Somewhat agree | 4
  Engaged or interested in the program: Somewhat disagree | 0
  Engaged or interested in the program: Completely disagree | 0
  Engaged or interested in the program: No response | 116
  Program helped learn about pneumonia & vaccination: Completely Agree | 110
  Program helped learn about pneumonia & vaccination: Somewhat agree | 26
  Program helped learn about pneumonia & vaccination: Somewhat disagree | 3
  Program helped learn about pneumonia & vaccination: Completely disagree | 0
  Program helped learn about pneumonia & vaccination: No response | 51

5. Secondary Outcome: Intervention Cost
Description: Measures PPPP intervention costs per participant. Consists of total program costs divided by number of participants. Value reported is the per-participant cost with measure type "number".
Time Frame: 3 months
Measure: Number; unit: $/participant
Arm/Group | PPPP Participants
Number analyzed (Participants) | 203
$/participant | 162.43

6. Secondary Outcome: Pharmacist Satisfaction
Description: Pharmacists who participated in the intervention were surveyed to determine their satisfaction with the program, including: 1) satisfaction with live action skit, 2) belief that PPPP was successful in educating participants, 3) belief that PPPP was successful in building trust in pharmacists among participants, 4) belief that PPPP was successful in increasing acceptance of pharmacists as immunizers, and 5) belief that PPPP will decrease barriers to vaccination among participants.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Pharmacy Staff: Pharmacy staff (pharmacy faculty and students) were surveyed after the completion of the program to determine their satisfaction with the program.
Arm/Group | Pharmacy Staff
Number analyzed (Participants) | 20
Participants
  Satisfaction with live action skit: Agree | 18
  Satisfaction with live action skit: Disagree | 1
  Satisfaction with live action skit: No response | 1
  Belief that PPPP successfully educated participnts: Agree | 19
  Belief that PPPP successfully educated participnts: Disagree | 1
  Belief that PPPP successfully educated participnts: No response | 0
  Belief that PPPP successfully built trust: Agree | 17
  Belief that PPPP successfully built trust: Disagree | 2
  Belief that PPPP successfully built trust: No response | 1
  Belief that PPPP successfully increased acceptance: Agree | 19
  Belief that PPPP successfully increased acceptance: Disagree | 1
  Belief that PPPP successfully increased acceptance: No response | 0
  Belief that PPPP decreased barriers to vaccination: Agree | 20
  Belief that PPPP decreased barriers to vaccination: Disagree | 0
  Belief that PPPP decreased barriers to vaccination: No response | 0

ADVERSE EVENTS:
Time Frame: Time of vaccination plus 7 days following receipt of vaccine
Description: Vaccine consent form stated risks & benefits of vaccine and instructed individuals suspecting an adverse event (AE) within 7 days post-vaccination to phone a 24-hour investigator hotline for immediate phone evaluation and determination of next steps. In the event of an AE, the VAERS reporting system form VAERS-1 (FDA) would have been utilized.
Groups:
- PPPP Participants - Vaccine Recipients: Subgroup of participants receiving the pneumococcal vaccine (Pneumococcal Vaccine Polyvalent (Pneumovax® 23))
Arm/Group | PPPP Participants - Vaccine Recipients
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less